CLINICAL TRIAL: NCT04060602
Title: Personalized Feedback Intervention to Reduce Risky Cannabis Use: Randomized Controlled Trial
Brief Title: Personalized Feedback Intervention to Reduce Risky Cannabis Use.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 143/2018
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Cannabis Use
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Feedback and Education (Experimental): This arm is provided personalized feedback concerning their cannabis use in addition to educational materials about risky cannabis use.
  Interventions: Behavioral: Personalized Feedback; Behavioral: Education
- Education (Active Comparator): This arm is provided educational materials about risky cannabis use.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Personalized Feedback — A report comparing the participant's cannabis use to peer usage, and summarizing problems experienced and risk associated with future use.
  Arms: Personalized Feedback and Education
Behavioral: Education — Canada's Lower-Risk Cannabis Use Guidelines prepared by the Centre for Addiction and Mental Health which outlines methods to help reduce health risks associated with cannabis use.

SUMMARY:
The purpose of this project is to determine whether participants who receive a personalized feedback report and educational materials about risky cannabis use will be less likely to report risky cannabis use at follow-up compared to participants who only received educational materials.

DETAILED DESCRIPTION:
This project aims to reduce risky cannabis use among those with less severe cannabis use, most of whom will never seek formal treatment. All of the participants will receive educational material regarding risky cannabis use and its prevention. Half of the participants will also be assigned by chance to receive a personalized feedback report.

The investigators hypothesize that:

1. Participants who receive the full personalized feedback intervention will be less likely to report risky cannabis use at 3- and 6-month follow-ups compared to participants who receive educational materials only (Primary Hypothesis).
2. Participants who receive the full personalized feedback intervention will report greater reductions in their perceptions of how much others use cannabis at a 3-month follow-up compared to participants who receive educational materials only.
3. Reductions in perceptions of how much others use cannabis at 3-month follow-up will be positively associated with reduction in the participant's risky cannabis use at 6-month follow-up.

A 2-arm parallel group randomized controlled trial will be conducted to test these hypotheses with follow-ups occurring at 3 and 6 months after randomization. Online media advertisements will be used to recruit people currently using cannabis. The advertisements will be placed across Canada using locations found successful in previous trials to rapidly recruit participants (e.g. Google AdWords).

ELIGIBILITY:
Inclusion Criteria:

* Score of 4 or more on the Alcohol, Smoking, and Substance Involvement Screening Test, Cannabis subscale (ASSIST)

Exclusion Criteria:

* Being under 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Cannabis Use in the last 30 days | 3 and 6 months
  Change in the number of days participant used cannabis in the past 30-days from baseline

SECONDARY OUTCOMES:
Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST, cannabis subscale) | Baseline, 3 and 6 months
  Change in cannabis subscale scores from baseline. Scores are calculated as a sum of six items and totals can range from 0 to 39 with higher scores indicating greater risk.
Perceptions of Cannabis Use by Peers in the past 3 months | Baseline, 3 months
  Change in participant's perceptions of how much their peers (same age and gender) use cannabis. Measured as a percentage of peers that do not use cannabis (%) and a 5-points Likert scale, 0 "Never" to 5 "Daily or Almost daily" of frequency of peer use

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham JA, Schell C, Bertholet N, Wardell JD, Quilty LC, Godinho A. Normative Misperceptions About Cannabis Use in a Sample of Risky Cannabis Users. Subst Abuse. 2023 Apr 6;17:11782218231166809. doi: 10.1177/11782218231166809. eCollection 2023. PMID 37051014
- See also: Description Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research